CLINICAL TRIAL: NCT06474806
Title: An Open-label, Two-part, Phase 2 Clinical Trial to Investigate the Safety and Diagnostic Performance of uPAR PET Imaging for Non-invasive Classification of ISUP Grades Among Patients With Localised, Untreated Prostate Cancer.
Brief Title: Safety and Diagnostic Performance of uPAR PET Imaging in Localised, Untreated Prostate Cancer
Acronym: uTRACE-101
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Curasight (Industry)
Collaborators: ABX CRO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 64Cu-DOTA-AE105-101; 2023-507111-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-06; First posted 2024-06-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial consist on 2 parts: Part 1 will evaluate 3 different doses of 64Cu-DOTA-AE105 in parallel (100, 150, or 200 MBq) in 27 patients (randomized 1:1:1) . Part 2 will evaluate 1 dose of 64Cu-DOTA-AE105 (200 MBq) in 141 patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100 MBq 64Cu-DOTA-AE105 (Experimental): For Part 1 of the trial, 9 patients will receive 100 MBq 64Cu-DOTA-AE105 Day 1 and Day 8
  Interventions: Drug: 64Cu-DOTA-AE105
- 150 MBq 64Cu-DOTA-AE105 (Experimental): For Part 1 of the trial, 9 patients will receive 150 MBq 64Cu-DOTA-AE105 Day 1 and Day 8
  Interventions: Drug: 64Cu-DOTA-AE105
- 200 MBq 64Cu-DOTA-AE105 (Experimental): For Part 1 of the trial, 9 patients will receive 200 MBq 64Cu-DOTA-AE105 Day 1 and Day 8.
  For Part 2 of the trial, additional 141 patients will receive 200 Mbq 64Cu-DOTA-AE105
  Interventions: Drug: 64Cu-DOTA-AE105

INTERVENTIONS:
Drug: 64Cu-DOTA-AE105 — AE105 is a uPAR-specific peptide that is bound to the chelator DOTA, which in turn holds the diagnostic radionuclide copper-64 (64Cu), which can be detected upon decay by PET imaging.

SUMMARY:
The goal of this clinical trial is to test if the experimental agent accurately determines the aggressiveness of prostate cancer (biopsy-verified ISUP grade). The aim is that the diagnostic PET imaging agent may be used as an alternative or supplement to biopsies in the monitoring of patients with low-risk prostate cancer in active surveillance.

Patients diagnosed with untreated, low-grade, localized prostate cancer may participate in the trial. The experimental diagnostic agent 64Cu-DOTA-AE105 is a radiopharmaceutical which is injected into the veins and binds to uPAR expressing cells in the tumour which can then be visualized in a PET scanner.

The main question the trial aims to answer is: Can the test drug be used alone or as a supplement to repeated biopsies to accurately assess the aggressiveness of prostate cancer?

The trial is divided in 2 parts:

* Participants in the first part will receive 2 injections of test drug on 2 different days.

  * The first day the participant will receive an injection of the test drug and then be asked to lie down in the PET/CT scanner so that images of the prostate can be taken. Before and after the injection/scanning procedure the participant will have tests done. These tests will include evaluation of health status, measurement of heart function by ECG plus blood and urine samples.
  * After 8 days the procedures, including injection of test drug and scanning, will be repeated.
* Participants in the second part of the trial will only have 1 injection of the test drug and subsequent PET/CT scanning. Like in Part 1 of the trial, tests will be done before and after the injection/ scanning procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pathology-verified prostate adenocarcinoma
* International Society of Urological Pathology (ISUP) grade 1 to 3
* Localised prostate cancer (N0 and M0 status) (only required for ISUP 3 patients)

  1. Newly diagnosed patients: Staging must be performed within 6 months from enrolment into the trial.
  2. Active surveillance: N0/M0 at the time of diagnosis and no clinical suspicion of prostate cancer outside the prostatic bed at the time of enrolment into the trial.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Prostate biopsy within 1 to 6 months (patients with a biopsy within the last month are excluded to avoid possible inflammation artefacts on the PET scan)

  1. The biopsy can be part of the primary staging, a confirmatory biopsy, or serial biopsy as part of an AS.
  2. At least 1 core must be MRI-guided.

Exclusion Criteria:

* Any prior treatment for prostate cancer (surgery, external beam radiation therapy, brachytherapy, hormone therapy, or chemotherapy)
* Chronic prostatitis (any signs or symptoms of chronic bacterial prostatitis or chronic pelvic prostatitis and pain syndrome, or known diagnosis of asymptomatic inflammatory prostatitis)
* Acute infections within the prostatic bed or lower urinary tract infections
* Participants have inadequate bone marrow, kidney, liver, heart, or lung function:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Standard uptake value (SUV) max at 30, 60, and 120 minutes post-injection (p.i.) - robustness | Day 1
  Part 1: mean of 3 independent readings of SUVmax at positron emission tomography (PET) aquisition times 30, 60, and 120 minutes p.1
Part 2: SUVmax at 60 minutes p.i. | 60 minutes post-injection
  Part 2: mean of 3 independent readings of SUVmax at PET aquisition time 60 minutes p.i.

SECONDARY OUTCOMES:
Part 1: SUVmax in PET acquisitions at 60 minutes p.i. | Day 1 and Day 8
  Part 1: mean of 3 independent readings of SUVmax at PET aquisition time 60 minutes Day 1 and Day 8
Part 1: Cmax from periodic radioactive counts from whole blood | Day 1
  Cmax from periodic radioactive counts from whole blood based on pre-injection and 5 post-injection samples
Part 1:Tmax from periodic radioactive counts from whole blood | Day 1
  Part 1: Tmax from periodic radioactive counts from whole blood based on pre-injection and 5 post-injection samples
Part 1: Area under curve (AUC) from periodic radioactive counts from whole blood | Day 1
  AUC from periodic radioactive counts from whole blood based on pre-injection and 5 post-injection samples
Part 1:Volume of distribution (Vd) from periodic radioactive counts from whole blood | Day 1
  Part 1: Vd from periodic radioactive counts from whole blood based on pre-injection and 5 post-injection samples
Part 1:Clearance from periodic radioactive counts from whole blood | Day 1
  Part 1: Clearance from periodic radioactive counts from whole blood based on pre-injection and 5 post-injection samples
Part 1: Elimination of 64Cu-DOTA-AE105 into a pooled urine sample | Day 1
  Part 1: Activity (MBq) per mL in urine samples pooled for the 3 hours following injection
Part 1: Inter-reader variability of SUVmax | Day 1
  Part 1: Variability of 3 independent SUVmax readings at 30, 60, and 120-minutes p.i.
Part 1:Intra-reader variability of SUVmax | Day 1
  Part 1: Variability of SUVmax readings at 30, 60, and 120-minutes p.i.
Part 1: Inter-reader variation in tumour visibility | Day 1
  Part 1: Tumor visibility in PET acquisitions evaluated by individual readings (numerical rating scale [NRS], 0-2 rating) at 30, 60, and 120 min p.i.
Part 1: Intra-reader variation in tumour visibility | Day 1
  Part 1: Tumor visibility in PET acquisitions evaluated by individual readings (numerical rating scale [NRS], 0-2 rating) at 30, 60, and 120 min p.i.
Part 1: SUVmax using different acquisition durations | Day 1
  Part 1: mean of 3 independent readings of SUVmax centered around 60 minutes p.i. in frame durations of 3-, 5-, 10-, 20-, 30-, and 40-minutes
Part 1: Variation in tumour visibility using different acquisition durations in the 200 MBq cohort | Day 1
  Part 1: median of 3 central readings of tumor visibility (NRS, 0-2 rating), centered around 60 minutes p.i. in frame durations of 3-, 5-, 10-, 20-, 30-, and 40-minutes
Part 2: SUVmax variation between local and central readers | 60 minutes post-injection
  Part 2: mean of 3 central readers and read of 1 local reader of SUVmax in PET acquisitions at 60 minutes p.i.
Part 2: Tumour visibility in PET acquisitions | 60 minutes post injection
  Part 2: median of 3 central readings of tumor visibility (NRS, 0-2 rating) and read of 1 local reader in PET acquisitions at 60 minutes p.i.
Part 2: Intra-reader variability of SUVmax | 60 minutes post injection
  Part 2: Variability of SUVmax readings at 60-minutes p.i.
Part 2: Inter-reader variability of SUVmax | 60 minutes post injection
  Part 2: Variability of 3 independent SUVmax readings at 60 minutes p.i.
Part 2: Inter-reader tumour visibility in PET acquisitions | 60 minutes post injection
  Part 2: individual readings by 3 central readers and 1 local reader of tumor visibility (NRS, 0-2 rating) in PET acquisitions at 60 minutes p.i.
Part 2: Intra-reader tumour visibility in PET acquisitions | 60 minutes post injection
  Part 2: individual readings by 3 central readers and 1 local reader of tumor visibility (NRS, 0-2 rating) in PET acquisitions at 60 minutes p.i.

OTHER OUTCOMES:
Incidence of adverse events | Day 3
  Part 2: Adverse events (AEs) will be assessed and graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, Study Director — Curasight
Locations (4):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Vejle Hospital, Vejle
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Skåne

IPD SHARING:
Plan to Share IPD: No